CLINICAL TRIAL: NCT03463915
Title: Randomized Controlled Trial Comparing Two Different Bladder Instillation Treatments for Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Clinical Trial Comparing Two Bladder Instillations for IC/BPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Olivia Cardenas-Trowers, M.D. (Other)
Responsible Party: Sponsor-Investigator, Olivia Cardenas-Trowers, M.D., Sponsor-Investigator, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18.0209
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Interstitial cystitis; Bladder pain syndrome; IC/BPS; Women; Pelvic pain; Urologic pain; Bladder instillation; Kenalog; Steroid
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain | interventions — Administration, Intravesical; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bladder instillation WITH triamcinolone acetonide (Active Comparator): Six weekly bladder instillations of standard cocktail plus triamcinolone acetonide. Standard cocktail= heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), and 0.5% bupivacaine (10 mL of 5 mg/mL) plus triamcinolone acetonide (1 vial, 40 milligrams (mg)/1 milliliters (mL).
  Interventions: Drug: Bladder instillation WITH triamcinolone acetonide
- Bladder instillation WITHOUT triamcinolone acetonide (Placebo Comparator): Six weekly bladder instillations of standard cocktail without triamcinolone acetonide. Standard cocktail= heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), and 0.5% bupivacaine (10 mL of 5 mg/mL).
  Interventions: Drug: Bladder instillation WITHOUT triamcinolone acetonide

INTERVENTIONS:
Drug: Bladder instillation WITH triamcinolone acetonide — Bladder instillation mixture of heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), 0.5% bupivacaine (10 mL of 5 mg/mL) plus triamcinolone acetonide (1 vial, 40 milligrams (mg)/1 milliliters (mL).
  Arms: Bladder instillation WITH triamcinolone acetonide
Drug: Bladder instillation WITHOUT triamcinolone acetonide — Bladder instillation mixture of heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), and 0.5% bupivacaine (10 mL of 5 mg/mL).
  Arms: Bladder instillation WITHOUT triamcinolone acetonide

SUMMARY:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a condition that results in long-term bladder and pelvic pain. IC/BPS affects women more often than men. How the disorder develops is not completely known. Bladder instillation is a commonly used treatment in which a mixture of different ingredients are passed into the bladder to help IC/BPS symptoms. There is room to learn more about bladder instillations and which ingredients in them work best. The purpose of this study is to compare the effectiveness of a bladder instillation that contains a steroid (triamcinolone acetonide) to a bladder instillation that does not contain a steroid to treat IC/BPS in women. The study hypothesis is that women with IC/BPS treated with bladder instillations that contain a steroid will have improved outcomes compared to women treated with bladder instillations that do not contain a steroid.

DETAILED DESCRIPTION:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a chronic pain disorder involving the genitourinary tract. IC/BPS disproportionately affects women with over 80% of patients with IC/BPS as female. Like other chronic pain conditions, IC/BPS is physically and emotionally taxing on patients. IC/BPS costs the United States over $100 million annually due to direct healthcare costs and loss of worker productivity. The exact pathophysiology of the disease is unknown, leading to a limitation in our ability to treat the disorder effectively. The current leading etiologic theory is that IC/BPS is a neurologically-derived chronic systemic pain syndrome due to its association with musculoskeletal pelvic pain, irritable bowel syndrome, chronic fatigue syndrome, fibromyalgia, and vulvodynia. Although several options exist to treat IC/BPS, therapeutic effects are often transient. Previous studies in chronic pain disorders have shown that multimodal treatment is more effective than single-agent treatment, so future therapy should aim to augment rather than replace current treatments. Bladder instillation is a commonly used treatment in which a mixture of different agents is instilled into the bladder to improve IC/BPS symptoms. The data on the efficacy of bladder instillations, as well as which ingredients in the mixture are effective, are limited. Small studies have shown the potential of steroids in decreasing IC/BPS; the mechanism of action is hypothesized to be due to decrease inflammation in the bladders of these patients. The knowledge gap that exists is the necessity of a steroid in the bladder instillation treatment for IC/BPS symptoms especially since this tends to be the most expensive ingredient.

To evaluate the utility of a steroid in the bladder instillation treatment of IC/BPS, we propose a randomized, double-blind, controlled trial that will compare the efficacy of bladder instillations with and without triamcinolone acetonide on IC/BPS symptoms in women. We hypothesize that the addition of triamcinolone acetonide in bladder instillation therapy will result in a more robust treatment response than bladder instillations without triamcinolone acetonide. Our rationale is based on 1) the results of small studies that showed improvement of IC/BPS symptoms with use of a steroid and 2) the hypothesized mechanism of action of steroids decreasing inflammation in the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older
* Women with IC/BPS who have a score of ≥ 6 on either index (problem or symptom index) of the O'Leary-Sant questionnaire who have selected bladder instillations as part of their IC/BPS treatment
* Suitability for follow-up

Exclusion Criteria:

* Contraindications and/or allergies to the ingredients used in the bladder instillations
* Diagnosis of idiopathic thrombocytopenic purpura
* Does not desire to undergo bladder instillation therapy or unwilling to undergo bladder instillation therapy on schedule mandated by study
* Have a known alternative diagnosis explaining bladder pain symptoms that would preclude the diagnosis of IC/BPS (e.g. radiation cystitis, active urinary tract infection with bacteria or fungus treated within last 2 weeks or diagnosed at index visit, bladder injury or trauma within the last 30 days)
* Inability to speak or read English
* Bladder instillation within the past 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Cardenas-Trowers, M.D., Principal Investigator — University of Louisville; Sean Francis, M.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Urogynecology at Springs Medical Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data and other supporting materials will be made available to approved investigators. Email requests to olivia.cardenas-trowers@louisville.edu.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 1 month and ending 24 months following article publication.
Access Criteria: Available to investigators whose proposed use of the data is for individual participant data meta-analysis and has been approved by an independent review committee for this purpose. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Clemens JQ, Meenan RT, Rosetti MC, Gao SY, Calhoun EA. Prevalence and incidence of interstitial cystitis in a managed care population. J Urol. 2005 Jan;173(1):98-102; discussion 102. doi: 10.1097/01.ju.0000146114.53828.82. PMID 15592041
- [Background] Nickel JC. Interstitial cystitis: a chronic pelvic pain syndrome. Med Clin North Am. 2004 Mar;88(2):467-81, xii. doi: 10.1016/S0025-7125(03)00151-2. PMID 15049588
- [Background] Aaron LA, Buchwald D. A review of the evidence for overlap among unexplained clinical conditions. Ann Intern Med. 2001 May 1;134(9 Pt 2):868-81. doi: 10.7326/0003-4819-134-9_part_2-200105011-00011. PMID 11346323
- [Background] Alagiri M, Chottiner S, Ratner V, Slade D, Hanno PM. Interstitial cystitis: unexplained associations with other chronic disease and pain syndromes. Urology. 1997 May;49(5A Suppl):52-7. doi: 10.1016/s0090-4295(99)80332-x. PMID 9146002
- [Background] Bullones Rodriguez MA, Afari N, Buchwald DS; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Urological Chronic Pelvic Pain. Evidence for overlap between urological and nonurological unexplained clinical conditions. J Urol. 2013 Jan;189(1 Suppl):S66-74. doi: 10.1016/j.juro.2012.11.019. PMID 23234637
- [Background] Clauw DJ, Schmidt M, Radulovic D, Singer A, Katz P, Bresette J. The relationship between fibromyalgia and interstitial cystitis. J Psychiatr Res. 1997 Jan-Feb;31(1):125-31. doi: 10.1016/s0022-3956(96)00051-9. PMID 9201654
- [Background] Dawson TE, Jamison J. Intravesical treatments for painful bladder syndrome/ interstitial cystitis. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006113. doi: 10.1002/14651858.CD006113.pub2. PMID 17943887
- [Background] Pazin C, de Souza Mitidieri AM, Silva AP, Gurian MB, Poli-Neto OB, Rosa-E-Silva JC. Treatment of bladder pain syndrome and interstitial cystitis: a systematic review. Int Urogynecol J. 2016 May;27(5):697-708. doi: 10.1007/s00192-015-2815-5. Epub 2015 Aug 14. PMID 26272202
- [Background] Chaparro LE, Wiffen PJ, Moore RA, Gilron I. Combination pharmacotherapy for the treatment of neuropathic pain in adults. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008943. doi: 10.1002/14651858.CD008943.pub2. PMID 22786518
- [Background] Cvach K, Rosamilia A. Review of intravesical therapies for bladder pain syndrome/interstitial cystitis. Transl Androl Urol. 2015 Dec;4(6):629-37. doi: 10.3978/j.issn.2223-4683.2015.10.07. PMID 26816864
- [Background] Barua JM, Arance I, Angulo JC, Riedl CR. A systematic review and meta-analysis on the efficacy of intravesical therapy for bladder pain syndrome/interstitial cystitis. Int Urogynecol J. 2016 Aug;27(8):1137-47. doi: 10.1007/s00192-015-2890-7. Epub 2015 Nov 20. PMID 26590137
- [Background] Soucy F, Gregoire M. Efficacy of prednisone for severe refractory ulcerative interstitial cystitis. J Urol. 2005 Mar;173(3):841-3; discussion 843. doi: 10.1097/01.ju.0000153612.14639.19. PMID 15711286
- [Background] Cox M, Klutke JJ, Klutke CG. Assessment of patient outcomes following submucosal injection of triamcinolone for treatment of Hunner's ulcer subtype interstitial cystitis. Can J Urol. 2009 Apr;16(2):4536-40. PMID 19364425
- [Derived] Cardenas-Trowers OO, Abraham AG, Dotson TK, Houlette BA, Gaskins JT, Francis SL. Bladder Instillations With Triamcinolone Acetonide for Interstitial Cystitis-Bladder Pain Syndrome: A Randomized Controlled Trial. Obstet Gynecol. 2021 May 1;137(5):810-819. doi: 10.1097/AOG.0000000000004348. PMID 33831942
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were women with IC/BPS who were recruited from January 2019 to October 2020 from the University of Louisville Female Pelvic Medicine & Reconstructive Surgery clinic in Louisville, KY.
Groups:
- Bladder Instillation WITH Triamcinolone Acetonide: Six weekly bladder instillations WITH triamcinolone acetonide: mixture of heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), 0.5% bupivacaine (10 mL of 5 mg/mL) plus triamcinolone acetonide (1 vial, 40 mg)/1 mL.
- Bladder Instillation WITHOUT Triamcinolone Acetonide: Six weekly bladder instillations WITHOUT triamcinolone acetonide: mixture of heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), and 0.5% bupivacaine (10 mL of 5 mg/mL).
Period: Overall Study
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Started | 45 | 45
Completed | 35 | 36
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Bladder Instillation WITH Triamcinolone Acetonide: Six weekly bladder instillations WITH triamcinolone acetonide: Bladder instillation mixture of heparin (10,000 units), 2% viscous lidocaine (10 mL), 8.4% sodium bicarbonate (15 mL of 1 mEq/mL), 0.5% bupivacaine (10 mL of 5 mg/mL) plus triamcinolone acetonide (1 vial, 40 mg/1 mL).
- Total: Total of all reporting groups
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.3) | 46.6 (14.0) | 42.0 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Treatment Response as Measured by the Total Score on the O'Leary-Sant Questionnaire
Description: Total scores range: 0-36 (0= no symptoms to 36= the most severe symptoms)
Time Frame: Assessed at baseline, 3 and 6 weeks; change from baseline to week 6 reported
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 45 | 45
scores on a scale | -6.7 (7.1) | -5.8 (8.0)

2. Secondary Outcome: Pelvic Pain and Urgency/Frequency (PUF) Questionnaire
Description: Total scores range: 0-35 (0= no symptoms to 35= the most severe symptoms)
Time Frame: Assessed at baseline, 3 and 6 weeks; change from baseline to week 6 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 33 | 36
score on a scale | -5.3 (5.1) | -2.7 (5.5)

3. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q)
Description: Total scores range: 0-100 (higher scores on the symptom-severity scale suggestive of greater severity of symptoms and higher scores on the quality-of-life scale suggestive of better quality of life)
Time Frame: Assessed at baseline, 3 and 6 weeks; change from baseline to week 6 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 34 | 34
score on a scale | -24.2 (19.1) | -18.8 (24.6)

4. Secondary Outcome: Pelvic Floor Distress Inventory (PFDI)
Description: 20 question self-administered questionnaire on the presence and absence of pelvic floor symptoms. Score ranges from 0 (least distress) to 300 (most distress).
Time Frame: Assessed at baseline, 3 and 6 weeks; change from baseline to week 6 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 29 | 29
score on a scale | -5.3 (9.5) | -6.4 (9.7)

5. Secondary Outcome: Sexual Function Measured by the Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) Questionnaire
Description: Measures sexual function in women with pelvic floor disorders. Queries about arousal, orgasm, partner-related issues, sexual quality, and desire. The tool also takes into account those who are not sexually active. The questionnaire was used in the study solely to determine if patients had improved dyspareunia (as a categorical variable).
Time Frame: Assessed at baseline, 3 and 6 weeks; change from baseline to week 6 reported
Measure: Number; unit: participants
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 36 | 40
participants | 4 | 4

6. Secondary Outcome: Change From Baseline in Treatment Response as Measured by the Visual Analogue Scale (VAS) for Pain
Description: VAS is measured on marking on a 10-centimeter (cm) ruler (measured in cm, 0= no pain and 10= most severe pain possible)
Time Frame: Assessed at baseline, 3 and 6 weeks; change from baseline to week 6 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 35 | 36
score on a scale | -1.9 (2.6) | -1.8 (2.4)

7. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: Adverse events will only be those determined to be related to the study drug
Time Frame: End of study (6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
Number analyzed (Participants) | 45 | 45
Participants | 1 | 5

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 weeks.
Description: The risk for these severe events is low because the risk of the intervention is known to be low.
Arm/Group | Bladder Instillation WITH Triamcinolone Acetonide | Bladder Instillation WITHOUT Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 5/45 | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bladder Instillation WITH Triamcinolone Acetonide (N=45) | Bladder Instillation WITHOUT Triamcinolone Acetonide (N=45)
Urethral pain (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Anxiety attack (Psychiatric disorders) | 1 (1) | 0 (0)
Strong bladder spasms (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03463915/Prot_SAP_000.pdf